CLINICAL TRIAL: NCT00953966
Title: Metabolic Changes Induced by Genetically Modified Potatoes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Professor J. Spranger, Charite University, Berlin, Germany
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: EA4/069/07
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Glucose Metabolism; Endocrine Metabolism; Satiety

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (7):
- Starch 1 (Other): Starch 1
  Interventions: Other: Genetically modified potatoes
- Starch 2 (Other): Starch 2
  Interventions: Other: Genetically modified potatoes
- Starch 3 (Other): Starch 3
  Interventions: Other: Genetically modified potatoes
- Starch 4 (Other): Starch 4
  Interventions: Other: Genetically modified potatoes
- Starch 5 (Other): Starch 5
  Interventions: Other: Genetically modified potatoes
- Starch 6 (Other): Starch 6
  Interventions: Other: Genetically modified potatoes
- Starch 7 (Other): Starch 7
  Interventions: Other: Genetically modified potatoes

INTERVENTIONS:
Other: Genetically modified potatoes — Starch from genetically modified potatoes

SUMMARY:
Starches from genetically modified potatoes, which differed in terms of amylose, amylopectin and phosphate content, were tested in a human randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* healthy males

Exclusion Criteria:

* no acute oder severe chronic diseases

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-06; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Glucose metabolism | 2 days

CONTACTS AND LOCATIONS:
Locations (1):
- Charité, Dept. of Endocrinology, Diabetes and Nutrition, Berlin, State of Berlin, Germany